CLINICAL TRIAL: NCT00212290
Title: Insulin Resistance and Central Nervous System (CNS) Function in Type 2 Diabetes
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DK61606 (completed)
Record Dates: First submitted 2005-09-20; First posted 2005-09-21 (Estimated); Last update posted 2010-02-15 (Estimated); Status verified 2010-02

CONDITIONS: Insulin Resistance; Type 2 Diabetes Mellitus
Keywords: impaired glucose tolerance
MeSH Terms: conditions — Insulin Resistance; Diabetes Mellitus, Type 2; Glucose Intolerance | interventions — Pioglitazone; Nateglinide

INTERVENTIONS:
Drug: pioglitazone
Drug: nateglinide
Drug: placebo

SUMMARY:
The purpose of this study is to examine the effects of treating insulin resistance on memory and attention, brain glucose utilization, and proteins in spinal fluid.

DETAILED DESCRIPTION:
Insulin resistant conditions such as impaired glucose tolerance, type 2 diabetes mellitus, and hyperinsulinemia have been associated with an increased risk for memory decline and for Alzheimer's disease. The main study will determine whether treatment with pioglitazone or nateglinide will improve verbal memory and selective attention for older adults with impaired glucose tolerance or mild type 2 diabetes. The main study will also characterize changes in blood concentrations of insulin, inflammatory markers, and the beta-amyloid peptides that are related to Alzheimer's disease. In one sub-study, participants will undergo brain positron emission tomography (PET) imaging before and after 16 weeks of treatment with pioglitazone, nateglinide, or placebo. The purpose of this sub-study is to determine the effects of treatment on brain glucose utilization. In a second sub-study, participants will undergo a lumbar puncture procedure before and after treatment. The purpose of this sub-study is to determine the effects of treatment on spinal fluid concentrations of insulin, inflammatory markers, and beta-amyloid peptides. Together these main and sub-studies should characterize the effects of insulin resistance on cognition and suggest a mechanism by which insulin resistant conditions increase risk for memory decline and for Alzheimer's disease.

ELIGIBILITY:
Inclusion Criteria:

* Impaired glucose tolerance OR mild type 2 diabetes mellitus OR normal blood sugar regulation
* Stable weight and activity level

Exclusion Criteria:

* Medications for diabetes
* Dementia
* Medications with known effects on memory
* Serious neurologic disease or head trauma
* Serious systemic illness (e.g., renal failure or uncontrolled hypertension)
* Serious psychiatric illness (e.g., schizophrenia or bipolar disorder)
* Allergy to pioglitazone or nateglinide

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2002-11; Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Verbal memory (main study)
Selective attention (main study)
Plasma beta-amyloid levels (main study)
Cerebral glucose metabolism (sub-study)
Inflammatory markers in spinal fluid (sub-study)
Beta-amyloid in spinal fluid (sub-study)

SECONDARY OUTCOMES:
Psychomotor speed
Verbal fluency
Blood levels of insulin, insulin degrading enzyme, cortisol and inflammatory markers

CONTACTS AND LOCATIONS:
Overall Officials: Suzanne Craft, PhD, Principal Investigator — VA Puget Sound Health Care System, University of Washington
Locations (2):
- United States (2):
  - VA Puget Sound Health Care System (Seattle Campus), Seattle, Washington
  - VA Puget Sound Health Care System (American Lake Campus), Tacoma, Washington